CLINICAL TRIAL: NCT04851405
Title: Implementing an Evidence-based Exercise Program to Reduce Falls in Community-dwelling Older Adults
Brief Title: Implementing an Evidence-based Exercise Program to Reduce Falls in Community-dwelling Older Adults (Otago)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Arthritis Research Centre of Canada (Other); Vancouver General Hospital (Other); Simon Fraser University (Other); Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Linda Li, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: H19-01760
Record Dates: First submitted 2021-04-09; First posted 2021-04-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Old Age; Debility; Fall
Keywords: Exercise; Strength Training; Fitbit
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Programme+ Intervention Group (OEP+) (Active Comparator): Physiotherapists receive OEP training, a 2 hour workshop on the coaching protocol using the OEP app, and online training on the Brief Action Plan Approach with 2 telephone practice sessions with an experienced Brief Action Plan counsellor.
  Each PT will deliver exercise program to 8 older adults. PTs will help older adults to set-up OEP app and Fitbit. PT will return bi-weekly over the course of two months (four visits total) for follow-up. During months 3-5, PTs will call participants three times times to review the exercise plan. The last visit will be an at-home visit which will occur 6 months after the initial visit. Between Months 7-12, PTs will continue to a phone call follow-up once a month to review the exercise routine.
  Older Adults will receive an OEP manual and cuff weights to be used with the strength training. They will also have access to the OEP app which allows the PT to prescribe exercises and record the participant's exercise goal.
  Interventions: Behavioral: Otago Exercise Programme+ (OEP+)
- Otago Exercise Programme Group (OEP) (Placebo Comparator): Physiotherapists receive OEP Training and a 2 hour workshop on just the counselling protocol.
  Each PT will deliver exercise program to 8 older adults. PTs will help older adults to set-up the Fitbit. For the first two months, PTs will provide bi-weekly home visits. During months 3-5, PTs will call participants three times times to review the exercise plan. The last visit will be an at-home visit which will occur 6 months after the initial visit.
  Older Adults will receive an OEP manual and cuff weights to be used with the strength training. They will also receive a Fitbit. Between Months 7-12, older adults will receive follow-up phone calls from the research staff.
  Interventions: Behavioral: Otago Exercise Programme (OEP)

INTERVENTIONS:
Behavioral: Otago Exercise Programme+ (OEP+) — Physiotherapists (PTs) will receive OEP and BAP training. They will provide at home visits and follow-up phone calls to the older adult participants (5 at home visits and 3 phone calls).
  Older adults will have access to the OEP app.
  Arms: Otago Exercise Programme+ Intervention Group (OEP+)
Behavioral: Otago Exercise Programme (OEP) — PTs will receive OEP training. They will provide at home visits and follow-up phone calls to the older adult participants (5 at home visits and 3 follow-up phone calls).
  Arms: Otago Exercise Programme Group (OEP)

SUMMARY:
Falls are a major health care problem for seniors. The Otago Exercise Program, which consists of strength and balance training delivered by a physiotherapist, can reduce falls in this population. We will test two methods to deliver the Otago program. These will include a new coaching approach by a physiotherapist with the use of a Fitbit to provide feedback versus the traditional delivery. The degree to which the program is delivered as intended by physiotherapists as well as the number of falls, risk of falling, and participation in walking activities in older adults will be assessed over 24 months. Lastly, we will assess if the coaching approach is a cost-effective option.

DETAILED DESCRIPTION:
Falls are a major health care problem for older adults (i.e., those aged ≥ 65 years) and health care systems. Falls account for 50% of injury-related admissions to hospital, 40% of admissions to nursing homes, and a 10% increase in home care services. They are also the leading cause of fatal injury among Canadians over 65 years old. This represents a significant health burden. Fortunately, falls are preventable. There is strong evidence that the Otago Exercise Program (OEP), physiotherapist (PT)-led home-based exercise program of strength and balance training, is effective at preventing falls in older adults with complex medical conditions. Originally developed in New Zealand the OEP has been implemented worldwide, but adherence to the program is a challenge. We propose that the suboptimal adherence is partly due to a lack of focus on behaviour change techniques such as self-monitoring and action planning in the delivery of OEP.

The investigators will use a mixed-methods approach, involving a RCT and in-depth interviews. The delivery of OEP+ vs OEP, from PTs, and its recipients, the older adults, will be determined at random. The training for the PT's will be provided by the Centre for Collaboration Motivation & Innovation (CCMI), a non-profit organization with a mandate to support the use of behaviour change techniques to improve health care. Prior to data collection, the PTs will attend a 2-hour workshop on the coaching protocol using the OEP app.

The goal of this project is to assess OEP+ as an implementation strategy to improve OEP delivery (by PTs) and adherence (by older adults).

ELIGIBILITY:
Inclusion Criteria (Older Adults):

* over 70 years of age
* self-report a non-syncopal fall corroborated by an informant, in the previous six months
* are able to walk three meters with or without an assistive device
* have a Mini-Mental State Examination score > 24/30
* have a Physiological Profile Assessment composite score of at least 1.0 standard deviation above age-normative value or have a Timed Up and Go test > 15 seconds, or had one additional non-syncopal fall in the previous 12 months
* live in an area served by Vancouver Coastal Health
* understand, speak, and read English proficiently
* have access to a mobile device
* are willing to have their OEP sessions audio-recorded
* able to provide written informed consent

Exclusion Criteria (Older Adults):

* people not meeting the criteria above

Inclusion Criteria (Physiotherapists):

* willing to participate in training on the OEP
* complete the BAP training
* be audio-recorded during the OEP sessions
* be randomized to the OEP group with coaching or without coaching

Exclusion Criteria (Physiotherapists):

* not willing to participate in the above criteria

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Physiotherapist-level outcome - Brief Action Planning (BAP) Scores | During the 12-month intervention
  This measure includes 33 items from three domains: 1) BAP content, 2) warmth and tone, and 3) overall interaction quality (total score: 0-35, higher score = better). The scores will be derived from the physiotherapists' sessions with the first, middle (Participant 3 or 4 out of 8) and last older adult participant. The recording from these treatment sessions will be coded and analysed by one of four researchers. The average of BAP scores of the middle and last participants for each PT will be used in the analysis .
Older Adult-Level Outcome - rate of adherence to the Otago Exercise Program (OEP) | During the 12-month intervention
  The number of exercise completed out of the total number of exercise prescribed during the intervention period

SECONDARY OUTCOMES:
Older Adult-Level Outcome - Number of Falls | During the 12-month intervention
  Number of falls reported by the older adult participants. We define falls as "an event which results in a person coming to rest inadvertently on the ground or floor or other lower level".
Older Adult-Level Outcome - Number of Falls | During the 12 months after the intervention (i.e., 13-24 months)
  Number of falls during the reported. We define falls as "an event which results in a person coming to rest inadvertently on the ground or floor or other lower level".
Older Adult-Level Outcome - Physiological Profile Assessment© (PPA) | Baseline
  PPA assesses risk of falls. Based on the performance of five domains (postural sway, hand reaction time, quadriceps strength, proprioception, and edge contrast sensitivity), a fall risk score will be computed for each participant. The PPA has a 75% predictive accuracy for falls in older people. A PPA z-score of 0-1 indicates mild risk, >1-2 indicates moderate risk, >2-3 indicates high risk, and >3 and above indicates marked risk.
Older Adult-Level Outcome - Physiological Profile Assessment© (PPA) | 6 months
  PPA assesses risk of falls. Based on the performance of five domains (postural sway, hand reaction time, quadriceps strength, proprioception, and edge contrast sensitivity), a fall risk score will be computed for each participant. The PPA has a 75% predictive accuracy for falls in older people. A PPA z-score of 0-1 indicates mild risk, >1-2 indicates moderate risk, >2-3 indicates high risk, and >3 and above indicates marked risk.
Older Adult-Level Outcome - Physiological Profile Assessment© (PPA) | 12 months
  PPA assesses risk of falls. Based on the performance of five domains (postural sway, hand reaction time, quadriceps strength, proprioception, and edge contrast sensitivity), a fall risk score will be computed for each participant. The PPA has a 75% predictive accuracy for falls in older people. A PPA z-score of 0-1 indicates mild risk, >1-2 indicates moderate risk, >2-3 indicates high risk, and >3 and above indicates marked risk.
Older Adult-Level Outcome - Physiological Profile Assessment© (PPA) | 18 months
  PPA assesses risk of falls. Based on the performance of five domains (postural sway, hand reaction time, quadriceps strength, proprioception, and edge contrast sensitivity), a fall risk score will be computed for each participant. The PPA has a 75% predictive accuracy for falls in older people. A PPA z-score of 0-1 indicates mild risk, >1-2 indicates moderate risk, >2-3 indicates high risk, and >3 and above indicates marked risk.
Older Adult-Level Outcome - Physiological Profile Assessment© (PPA) | 24 months
  PPA assesses risk of falls. Based on the performance of five domains (postural sway, hand reaction time, quadriceps strength, proprioception, and edge contrast sensitivity), a fall risk score will be computed for each participant. The PPA has a 75% predictive accuracy for falls in older people. A PPA z-score of 0-1 indicates mild risk, >1-2 indicates moderate risk, >2-3 indicates high risk, and >3 and above indicates marked risk.
Older Adult-Level Outcome - Average Daily Step Count | Baseline
  Measured by averaging the daily step counts, recorded by a Fitbit worn at the ankle (the non-dominant side), over seven days.
Older Adult-Level Outcome - Average Daily Step Count | 6 months
  Measured by averaging the daily step counts, recorded by a Fitbit worn at the ankle (the non-dominant side), over seven days.
Older Adult-Level Outcome - Average Daily Step Count | 12 months
  Measured by averaging the daily step counts, recorded by a Fitbit worn at the ankle (the non-dominant side), over seven days.
Older Adult-Level Outcome - Average Daily Step Count | 18 months
  Measured by averaging the daily step counts, recorded by a Fitbit worn at the ankle (the non-dominant side), over seven days.
Older Adult-Level Outcome - Average Daily Step Count | 24 months
  Measured by averaging the daily step counts, recorded by a Fitbit worn at the ankle (the non-dominant side), over seven days.
Older Adult-Level Outcome - EuroQol-5D-5 Level version (EQ-5D-5L) | Baseline
  EQ-5D-5L is a generic preference-based utility measure composed of 5 domains of health (mobility, self-care, usual activities, pain, and anxiety/depression). Each domain contains 5 levels, with a '1' indicating no problem and a '5' indicating major problem. The 5 dimensions (i.e., the health state profile) will be converted into a weighted health state utility values between '0' and '1', where '1' represents "perfect health" and '0' represents a health state equivalent to death. Values less than '0' indicate a health state worse than death. These health state utility values will provide weightings for QALYs. We will employ Canadian conversion tariffs for transforming health state profiles into utility scores.
Older Adult-Level Outcome - EuroQol-5D-5 Level version (EQ-5D-5L) | 6 months
  EQ-5D-5L is a generic preference-based utility measure composed of 5 domains of health (mobility, self-care, usual activities, pain, and anxiety/depression). Each domain contains 5 levels, with a '1' indicating no problem and a '5' indicating major problem. The 5 dimensions (i.e., the health state profile) will be converted into a weighted health state utility values between '0' and '1', where '1' represents "perfect health" and '0' represents a health state equivalent to death. Values less than '0' indicate a health state worse than death. These health state utility values will provide weightings for QALYs. We will employ Canadian conversion tariffs for transforming health state profiles into utility scores.
Older Adult-Level Outcome - EuroQol-5D-5 Level version (EQ-5D-5L) | 12 months
  EQ-5D-5L is a generic preference-based utility measure composed of 5 domains of health (mobility, self-care, usual activities, pain, and anxiety/depression). Each domain contains 5 levels, with a '1' indicating no problem and a '5' indicating major problem. The 5 dimensions (i.e., the health state profile) will be converted into a weighted health state utility values between '0' and '1', where '1' represents "perfect health" and '0' represents a health state equivalent to death. Values less than '0' indicate a health state worse than death. These health state utility values will provide weightings for QALYs. We will employ Canadian conversion tariffs for transforming health state profiles into utility scores.
Older Adult-Level Outcome - EuroQol-5D-5 Level version (EQ-5D-5L) | 18 months
  EQ-5D-5L is a generic preference-based utility measure composed of 5 domains of health (mobility, self-care, usual activities, pain, and anxiety/depression). Each domain contains 5 levels, with a '1' indicating no problem and a '5' indicating major problem. The 5 dimensions (i.e., the health state profile) will be converted into a weighted health state utility values between '0' and '1', where '1' represents "perfect health" and '0' represents a health state equivalent to death. Values less than '0' indicate a health state worse than death. These health state utility values will provide weightings for QALYs. We will employ Canadian conversion tariffs for transforming health state profiles into utility scores.
Older Adult-Level Outcome - EuroQol-5D-5 Level version (EQ-5D-5L) | 24 months
  EQ-5D-5L is a generic preference-based utility measure composed of 5 domains of health (mobility, self-care, usual activities, pain, and anxiety/depression). Each domain contains 5 levels, with a '1' indicating no problem and a '5' indicating major problem. The 5 dimensions (i.e., the health state profile) will be converted into a weighted health state utility values between '0' and '1', where '1' represents "perfect health" and '0' represents a health state equivalent to death. Values less than '0' indicate a health state worse than death. These health state utility values will provide weightings for QALYs. We will employ Canadian conversion tariffs for transforming health state profiles into utility scores.
Older Adult-Level Outcome - Health Resource Utilization Questionnaire (HRU) | Baseline
  The HRU asks for specific details regarding health professional visits, admissions to hospital, laboratory tests, use of medications, purchase of adaptive aids, and the productivity loss incurred by the older adults and their caregivers due to the person's poor health
Older Adult-Level Outcome - Health Resource Utilization Questionnaire (HRU) | 3 months
  The HRU asks for specific details regarding health professional visits, admissions to hospital, laboratory tests, use of medications, purchase of adaptive aids, and the productivity loss incurred by the older adults and their caregivers due to the person's poor health
Older Adult-Level Outcome - Health Resource Utilization Questionnaire (HRU) | 6 months
  The HRU asks for specific details regarding health professional visits, admissions to hospital, laboratory tests, use of medications, purchase of adaptive aids, and the productivity loss incurred by the older adults and their caregivers due to the person's poor health
Older Adult-Level Outcome - Health Resource Utilization Questionnaire (HRU) | 9 months
  The HRU asks for specific details regarding health professional visits, admissions to hospital, laboratory tests, use of medications, purchase of adaptive aids, and the productivity loss incurred by the older adults and their caregivers due to the person's poor health
Older Adult-Level Outcome - Health Resource Utilization Questionnaire (HRU) | 12 months
  The HRU asks for specific details regarding health professional visits, admissions to hospital, laboratory tests, use of medications, purchase of adaptive aids, and the productivity loss incurred by the older adults and their caregivers due to the person's poor health

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — Professor
Locations (1):
- Arthritis Research Canada, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No